CLINICAL TRIAL: NCT02563873
Title: Bowditch Revisited: Defining the Optimum Heart Rate Range in Chronic Heart Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Leeds (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Principal Investigator, John Gierula, NIHR Fellow and Cardiac Physiologist, University of Leeds
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 12/YH/0097
Record Dates: First submitted 2015-07-22; First posted 2015-09-30 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-05

CONDITIONS: Chronic Heart Failure

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard pacemaker settings (No Intervention): Standard pacemaker settings will be programmed and the patient will complete a symptom limited exercise tolerance test with metabolic gas exchange
- Tailored pacemaker settings (Experimental): The pacemaker settings will be altered to match optimal heart rate range with respect to cardiac contractility, as determined by echocardiography. This will be programmed and the patient will complete a symptom limited exercise tolerance test with metabolic gas exchange.
  Interventions: Device: Tailored pacemaker settings

INTERVENTIONS:
Device: Tailored pacemaker settings — Tailored pacemaker settings, optimised for cardiac contractility: Pacemaker settings, optimised for cardiac contractility as determined by echocardiography, will be programmed
  Arms: Tailored pacemaker settings

SUMMARY:
The investigators are examining the relationship between heart rate and heart contraction in patients with heart failure and pacemakers, aiming to improve quality of life.

DETAILED DESCRIPTION:
Heart rate lowering is a cornerstone of the management of chronic heart failure (CHF) and the degree of lowering is closely related to improvements in longevity, hospitalisation rate and heart function. The investigators have shown that increasing heart rates using pacemakers does not increase exercise capacity in CHF patients. This might be because the optimal heart rate range for contraction is narrower for patients with CHF. At higher heart rates, heart contraction might be less strong. The investigators now want to examine the relationship between heart rate and heart contraction in patients with heart failure and pacemakers. Tailored pacemaker heart rate setting's, individually optimised for heart contractility as assessed by cardiac ultrasound, will be investigated to examine the effects on exercise tolerance .

ELIGIBILITY:
Inclusion Criteria:

* stable CHF
* Cardiac Resynchronisation Therapy (CRT) device for >3 months,
* able to walk on treadmill

Exclusion Criteria:

* unable to walk on treadmill,
* unstable angina pectoris
* uncontrolled heart rate
* prescribed calcium channel blocker
* significant aortic stenosis
* significant airways disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2015-10; Primary Completion 2017-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Change in Exercise Time | Assessed following the second treadmill test, 1 week later
  Exercise duration in seconds

SECONDARY OUTCOMES:
Change in Peak Oxygen Consumption (pVO2) | Assessed following the second treadmill test, 1 week later
  Peak Oxygen Consumption (pVO2) measured by metabolic gas exchange

CONTACTS AND LOCATIONS:
Overall Officials: John Gierula, BSc, Principal Investigator — University of Leeds
Locations (1):
- Leeds Institute of Cardiovascular and Metabolic Medicine, Leeds, West Yorkshire, United Kingdom

REFERENCES:
- [Background] Al-Najjar Y, Witte KK, Clark AL. Chronotropic incompetence and survival in chronic heart failure. Int J Cardiol. 2012 May 17;157(1):48-52. doi: 10.1016/j.ijcard.2010.11.018. Epub 2010 Dec 23. PMID 21185094
- [Background] Shelton RJ, Ingle L, Rigby AS, Witte KK, Cleland JG, Clark AL. Cardiac output does not limit submaximal exercise capacity in patients with chronic heart failure. Eur J Heart Fail. 2010 Sep;12(9):983-9. doi: 10.1093/eurjhf/hfq086. Epub 2010 Jun 4. PMID 20525704
- [Background] Witte KK, Clark AL. Chronotropic incompetence does not contribute to submaximal exercise limitation in patients with chronic heart failure. Int J Cardiol. 2009 May 29;134(3):342-4. doi: 10.1016/j.ijcard.2008.02.014. Epub 2008 Jun 20. PMID 18571253
- [Background] Thackray SD, Ghosh JM, Wright GA, Witte KK, Nikitin NP, Kaye GC, Clark AL, Tweddel A, Cleland JG. The effect of altering heart rate on ventricular function in patients with heart failure treated with beta-blockers. Am Heart J. 2006 Oct;152(4):713.e9-13. doi: 10.1016/j.ahj.2006.07.007. PMID 16996845
- [Background] Witte KK, Clark AL. Resting left ventricular function, however measured, is poorly related to exercise capacity in chronic heart failure. Am J Cardiol. 2006 Sep 1;98(5):709-10. doi: 10.1016/j.amjcard.2006.05.002. Epub 2006 Jul 5. No abstract available. PMID 16923470
- [Background] Witte KK, Clark AL. Chronotropic incompetence in heart failure. J Am Coll Cardiol. 2006 Aug 1;48(3):595; author reply 595-6. doi: 10.1016/j.jacc.2006.05.014. Epub 2006 Jul 12. No abstract available. PMID 16875998
- [Background] Witte KK, Cleland JG, Clark AL. Chronic heart failure, chronotropic incompetence, and the effects of beta blockade. Heart. 2006 Apr;92(4):481-6. doi: 10.1136/hrt.2004.058073. Epub 2005 Sep 13. PMID 16159968
- [Background] Thackray SD, Witte KK, Nikitin NP, Clark AL, Kaye GC, Cleland JG. The prevalence of heart failure and asymptomatic left ventricular systolic dysfunction in a typical regional pacemaker population. Eur Heart J. 2003 Jun;24(12):1143-52. doi: 10.1016/s0195-668x(03)00199-4. PMID 12804929
- [Derived] Gierula J, Paton MF, Lowry JE, Jamil HA, Byrom R, Drozd M, Garnham JO, Cubbon RM, Cairns DA, Kearney MT, Witte KK. Rate-Response Programming Tailored to the Force-Frequency Relationship Improves Exercise Tolerance in Chronic Heart Failure. JACC Heart Fail. 2018 Feb;6(2):105-113. doi: 10.1016/j.jchf.2017.09.018. Epub 2017 Dec 6. PMID 29226818